CLINICAL TRIAL: NCT06883994
Title: Fermented Vegetables and Gut Microbiome Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bess L Caswell, Research Nutritionist, USDA, Western Human Nutrition Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FL125; USDA 2032-10700-002-000D (Other Grant/Funding Number: US Department of Agriculture (USDA) Agricultural Research Service (ARS))
Record Dates: First submitted 2025-03-10; First posted 2025-03-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-09

CONDITIONS: Fermented Vegetable Intake; Fermented Vegetable Acceptability; Gut Health; Gut Microbiome; Gastrointestinal Immune Function; Microbiome
Keywords: Fermented vegetables; Fermented foods; Nutrition; Adults; Immune function; Gastrointestinal (GI) health; Gut microbiome; GI tract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fermented vegetable consumption (Experimental): Participants will complete a 1-week baseline with no fermented food intake, followed by a 4-day fermented vegetable intervention, and then a 1-week follow-up period with no fermented food intake.
  Interventions: Other: Fermented vegetable intervention

INTERVENTIONS:
Other: Fermented vegetable intervention — Participants will be provided with reduced-sodium fermented vegetables developed by Dr. Ilenys Pérez-Díaz at the USDA-ARS Food Science and Market Quality and Handling Research Unit. The fermented, refrigerated vegetables have been shown to have Lactiplantibacillus spp. content >10^7 CFU/mL at 21 days shelf-life.
  Products are prepared in a Good Manufacturing Practices Facility at North Carolina State University, Department of Food, Bioprocessing, and Nutrition Sciences.
  The fermented vegetables will be shipped in coolers on cold packs with temperature indicators to the WHNRC. Participants will be asked to consume two pre-packaged 50g servings of fermented vegetables a day, for a total daily serving of 100g, not to heat the fermented vegetables prior to consumption, to log their consumption and to rate the acceptability of the fermented vegetables. They will be advised to avoid other fermented foods and to otherwise maintain their habitual diet.

SUMMARY:
The purpose of this research is to determine the effect of fermented vegetable consumption on LAB abundance and tolerability of the intervention in young healthy people before conducting a full RCT with older participants.

DETAILED DESCRIPTION:
The purpose of this research is to determine the tolerability of fermented vegetable consumption and its effect on lactic acid bacteria (LAB) abundance in healthy people. There is evidence from previous studies that eating fermented foods containing live microbes can affect the gut microbiome and gut health, but there is little information on the impact of fermented vegetables, specifically.

This research will expand the limited existing literature on the effect of fermented vegetable intake on LAB abundance, GI symptoms, fecal consistency and frequency.

Specific knowledge will be produced regarding the magnitude and variation in the increase in LAB bacterial load during fermented vegetable consumption and whether one week is sufficient for LAB to pass out of the gastrointestinal tract. The effect of fermented vegetable consumption on total salivary sIgA levels in healthy adults will also be determined.

The study will also produce knowledge on whether symptoms of bloating and flatulence will improve with fermented vegetables. Stool consistency, stool frequency, GI symptoms, blood pressure and product acceptability data will inform the study design for a future randomized controlled trial of the effects of fermented vegetables on gut microbiome composition and function, gut health and immune function.

The impacts of fermented vegetable consumption on the human gut microbiome, intestinal permeability, and GI inflammation will also be determined with in vitro experiments.

ELIGIBILITY:
We will enroll non-obese adults aged 18-65 years, with BMI between 18.5 and 39.9 kg/m2. We will exclude people with a high blood pressure, who cannot consume fermented vegetables, and those among whom a medical condition, use of medication, use of probiotic supplements or consumption of fermented foods may influence trial outcomes. Those who are uncomfortable with the stool sample collection protocol, or who may not be able to complete the stool samples due to infrequent bowel movements, will also be excluded.

Adults who are unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant women, and prisoners will be excluded from participation in the study.

Inclusion Criteria:

* Age 18 - 65 years
* BMI 18.5 - 39.9 kg/m2

Exclusion Criteria:

* BMI less than 18.5 or greater than 39.9
* Pregnant or breastfeeding
* Allergy or sensitivity to any fruit or vegetable
* Dietary restriction preventing consumption of fermented vegetables
* Consumption of probiotic supplements, foods or drinks in the past month

  * Probiotic supplements include any tablets, liquids, powders, chewables or other formulations that provide high-quantity, live probiotic microbes
  * Probiotic foods and drinks include products labeled as 'probiotic' because they contain live microbes in types and quantities that may confer a health benefit
* Regular consumption, defined as consumption more than once per week in the past two weeks, of live microbe-containing fermented vegetables or cultured dairy products, such as kimchi, refrigerated fermented pickles, traditional (lacto-fermented) sauerkraut, yogurt, or kefir

  * In case of less frequent consumption, defer study start such that baseline assessments are completed at least two weeks after last intake
* Unwillingness to abstain from non-study fermented foods and probiotics during the trial
* Uncomfortable with or unwilling to complete stool sample or saliva collections
* Current participation in another interventional research study
* Having fewer than 3 bowel movements per week
* Unmanaged hypertension, defined as blood pressure greater than or equal to 140/90 mmHg
* Current diagnosis of:

  * Disease that affects the immune system or causes immune impairment, including HIV/AIDS
  * Cancer
  * Diabetes
  * Asthma with daily medication
  * Primary immune deficiency
  * Auto-immune disease
  * Chronic gastrointestinal disorder (e.g. Crohn's disease, irritable bowel syndrome, colitis, gastric ulcer)
  * Chronic kidney disease
* Current use for 2 weeks or longer of:

  * Any drug that affects the immune system, such as immunosuppressants, immune modifying drugs, or corticosteroids (e.g. cortisone, prednisone, methylprednisolone)
  * Biologics (e.g. Lantus, Remicade, Rituxan, Humira, Herceptin, Avastin, Lucentis, Enbrel)
  * GLP-1 agonists, such as semaglutide and tirzepatide.
  * Antidiabetic medications, such as Metformin.
  * Diuretics, such as Hydrochlorothiazide
* Use of sulfonamides or antimicrobials, including antibiotics, antifungals, antivirals, and antiparasitic medications in the past 3 months
* Use of laxatives in the past 2 weeks
* Currently undergoing cancer treatment with radiation or drugs
* History of gastrointestinal surgery that would impact study outcomes, such as gastric bypass, intestinal resection, surgeries of the liver or pancreas, or removal of part or all of any organ of the GI tract
* Having within the past 2 weeks:

  * Diarrheal illness, defined as passing 3 or more abnormally loose or watery stools in a 24-hour period
  * Persistent vomiting
  * Fever
* Having within the past 3 months:

  * Surgery
  * Hospitalization
* Having within the past 1 month:

  * Colonoscopy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Lactic acid bacteria (LAB) cell count in stool | At the end of 1-week un-intervened baseline, 4-day intervention and 1-week un-intervened follow-up.
  Bacterial DNA extracted from subject stools will be used for quantitative polymerase chain reaction (qPCR) analysis using primers specific for lactic acid bacteria (LAB) in the intervention food, to estimate bacterial cell count per gram of wet stool.

SECONDARY OUTCOMES:
GI symptoms | At the end of 1-week un-intervened baseline, 4-day intervention and 1-week un-intervened follow-up.
  GI symptoms will be measured using a 10-symptom health questionnaire with degree of discomfort ranked in one of four categories: absent, mild, moderate or severe.
Stool frequency | Throughout 1-week un-intervened baseline, 4-day intervention and 1-week un-intervened follow-up.
  Stool frequency will be measured by self-report in stool diaries and summarized by number of bowel movements per day within each study phase.
Stool consistency | Throughout 1-week un-intervened baseline, 4-day intervention and 1-week un-intervened follow-up.
  Stool consistency will be measured by self-report in stool diaries, with stool consistency being classified into 1 of 7 categories according to the Bristol Stool Scale.
Salivary secretory immunoglobulin A | At the end of 1-week un-intervened baseline, 4-day intervention and 1-week un-intervened follow-up.
  Total salivary secretory immunoglobulin A (sIgA) will be extracted then measured in duplicate by enzyme-linked immunosorbent assay (ELISA)

OTHER OUTCOMES:
Acceptability of fermented vegetables | Throughout 4-day intervention period
  Acceptability of fermented vegetables will be described by participant rating of the appearance, aroma/smell, taste, texture and overall acceptability of the food on a scale of 1 (worst) to 10 (best).
Blood pressure | At the end of 1-week un-intervened baseline, 4-day intervention and 1-week un-intervened follow-up.
  Blood pressure will be measured using an automated vital signs monitor with blood pressure cuff.
Gut microbiome composition | At the end of 1-week un-intervened baseline
  Stool samples collected at the end of 1-wk baseline will be cultured for 48hr in batch fermentations with digested, pureed vegetables and fermented vegetables will be collected at the 0hr, 4hr, 24hr, 48hr timepoints and used for 16S ribosomal ribonucleic acid (rRNA) analysis.
Intestinal permeability | At the end of 1-week un-intervened baseline, 4-day intervention and 1-week un-intervened follow-up.
  Samples collected from batch fermentations will be applied to an in vitro gut barrier model consisting of Caco-2 cells. Transepithelial electrical resistance (TEER) will be used to evaluate intestinal permeability.
Gastrointestinal inflammation | At the end of 1-week un-intervened baseline, 4-day intervention and 1-week un-intervened follow-up.
  Gut inflammation will be assessed by measuring molecules in stool and/or the response of intestinal epithelial cell cultures to fecal waters from a single stool sample.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle G Lemay, PhD, Principal Investigator — USDA, Western Human Nutrition Research Center; Bess L Caswell, PhD, Principal Investigator — USDA, Western Human Nutrition Research Center; Mary E Kable, PhD, Principal Investigator — USDA, Western Human Nutrition Research Center
Locations (1):
- USDA Western Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared at the time of study publication in accordance with USDA policy.
Time Frame: At the time of study publication, de-identified IPD will be permanently archived on a publicly assessible platform.
Access Criteria: De-identified IPD and supporting information will be publicly available.

DOCUMENTS (1):
  • Informed Consent Form (2025-04-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT06883994/ICF_000.pdf